CLINICAL TRIAL: NCT03914729
Title: Multicenter Randomized Controlled Trial of Mobilized Gluteus Maximus Muscle Fascia Flap Versus Primary Closure in the Treatment of Primary and Recurrent Pilonidal Sinus Disease.
Brief Title: GLUtEus Maximus Fascia Plasty Flap for Pilonidal Sinus
Acronym: GLUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199323
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal sinus; plasty; gluteus muscle fascia; ano-coccygeal plasty
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, parallel-arm randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Closure (Active Comparator): After pilonidal sinus is excised, subcutaneous fat and skin are closed in midline with a running suture
  Interventions: Procedure: Primary Closure
- Gluteus Maximus Plasty Flap (Active Comparator): After pilonidal sinus is excised, gluteus maximus fascia flaps will be mobilised, approximated in the midline and fixed with a running suture. Subcutaneous fat and skin are closed in midline with a running suture.
  Interventions: Procedure: Gluteus Maximus Fascia Plasty Flap

INTERVENTIONS:
Procedure: Primary Closure — A symmetrical elliptical incision of skin and subcutaneous fat around primary and secondary orifices is performed. The cyst is excised en bloc down to the sacral fascia and removed. The lateral edges of the wound are approximated and sutured in the midline: subcutaneous fat - with a running suture, skin - with a separate running suture.
  Arms: Primary Closure
Procedure: Gluteus Maximus Fascia Plasty Flap — A symmetrical elliptical incision of skin and subcutaneous fat around primary and secondary orifices is performed. The cyst is excised en bloc down to the sacral fascia and removed. The lateral edges of the gluteus maximus muscles fascia bilaterally are mobilised in the direction from the fixation point to the sacrum and for 3-4 cm in lateral direction. The fascia flaps edges are approximated and fixed in the midline with a running suture. The subcutaneous fat is closed with a running suture, skin is closed with a separate running suture.
  Arms: Gluteus Maximus Plasty Flap

SUMMARY:
Surgical treatment is still gold standard for pilonidal sinus disease. Several surgical techniques have been proposed to treat this disease in the last two decades. A new method - midline excision of pilonidal sinus and wound closure using gluteus maximus fascia plasty flap (GMFF) - was proposed recently as a new method of treatment that results in low reccurence rate and good cosmetic results.

The aim of this study is to compare a new method (GMFF) with a traditional method (midline excision and primary closure) in terms of recurrence rate, complications and patient satisfaction with results.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is a rather rare benign condition (about 26 cases per 100,000 population) that affects primarily young adults. Because of purulent nature it is treated with surgery only.

Traditional surgical techniques encompass midline excision of the purulent cyst and either leaving the wound "lay open" for secondary closure or midline primary closure. The latter method has a major drawback of high recurrence rate and very long healing and patient disability periods. Therefore alternative techniques to close the wound after pilonidal sinus excision were proposed. In some a muscular-cutaneous flaps are created and the wound is closed in a Z- or Y- or other shape manner. The recurrence rate of these techniques is significantly lower than with a traditional midline closure, but healing time and final cosmetic results are far from ideal in patient view.

Recently a new method of wound closure was developed independently by a few groups that includes bilateral mobilisation of gluteus maximus muscles fascia and midline closure of the wound. Preliminary results demonstrated that this method leads to lower recurrence rate and better cosmetic results because the natal cleft is saved.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Chronic primary or recurrent pilonidal sinus at the remission stage.
3. Presence or absence of secondary orifices.
4. Planned surgical treatment with excision of pilonidal sinus.
5. Location of secondary orifices less than 2 cm from the natal cleft.
6. The distance between bilateral symmetrical secondary orifices less than 2 cm.
7. American Society Anesthesiologists (ASA) score 1 to 3

Non-inclusion Criteria:

1. Acute pilonidal sinus abscess.
2. The secondary openings (orifice) position more than 2 cm from the midline.
3. ASA 4-5.
4. Predictable impossibility of following the protocol.
5. Pregnancy

Exclusion criteria:

1 The patients lost for the further observation. 2. The patient's refusal to continue participate in the investigation.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | starting from 6 months after surgery and up to 5 years after surgery
  The rate of disease recurrence (clinical picture of pilonidal sinus and/or appearance of new openings in the intergluteal cleft and/or chronic unhealing wound and/or residual cavity in the wound area as confirmed by the soft tissue ultrasound)

SECONDARY OUTCOMES:
Operative time | 1 day
  The length of surgery in minutes
Bloodloss | 1 day
  The amount of blood lost during surgery
Postoperative pain intensity - early postoperative period | On 1st, 3rd, 5th and 7th postoperative day
  Pain intensity will be evaluated twice a day (in the morning and in the evening) with a patient-reported Visual Analog Scale (VAS) that ranges from 0 to 10 with 0 representing no pain and 10 representing intolerable pain. A total score will be recorded.
Postoperative pain intensity - late postoperative period | On 10th, 14th, 21st, 30 day after surgery
  Pain intensity will be evaluated once a day with a patient-reported Visual Analog Scale (VAS) that ranges from 0 to 10 with 0 representing no pain and 10 representing intolerable pain. A total score will be recorded.
Surgical site infection rate | 3 month after surgery
  The rate of infectious inflammation of the wound as confirmed by the observing doctor
Inhospital stay | 30 days
  The duration of treatment after surgery untill discharge from the hospital (in days)
Wound hemorrhage rate | Within 30 days from surgery
  The rate of hemorrhage from wound edges
Wound seroma rate | 90 days after surgery
  The rate of seroma detection in the wound area as confirmed by soft tissues ultrasound
Wound healing rate | 6 months after surgery
  The proportion of patients having their wound completely healed
Wound healing speed | 5 years after surgery
  The time period between surgery and complete healing of the wound
Secondary surgery rate | 5 years
  The rate of surgical procedures after initial surgery performed for recurrent disease and/or wound complications
Patient satisfaction with cosmetic results | 6 months, 1 year, 3 years, 5 years after surgery
  Patient-reported with a scale 0-10, where 0 corresponds to "completely unsatisfactory" and 10 corresponds to "completely satisfactory". A total score is registered.
Overall quality of life | 1-7 days before surgery, 1 month, 3 months, 1 year, 3 years, 5 years after surgery
  Assessed with patient-reported questionnaire SF-36. A total score in each of 8 sections will be calculated and transformed into a 0-100 scale with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disability

CONTACTS AND LOCATIONS:
Overall Officials: Inna Tulina, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University; Petr Tsarkov, Prof., Study Director — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally Invasive Surgery - I.M. Sechenov First Moscow State Medical University, Moscow, Russia

REFERENCES:
- [Result] Chintapatla S, Safarani N, Kumar S, Haboubi N. Sacrococcygeal pilonidal sinus: historical review, pathological insight and surgical options. Tech Coloproctol. 2003 Apr;7(1):3-8. doi: 10.1007/s101510300001. PMID 12750948
- [Result] Sondenaa K, Andersen E, Nesvik I, Soreide JA. Patient characteristics and symptoms in chronic pilonidal sinus disease. Int J Colorectal Dis. 1995;10(1):39-42. doi: 10.1007/BF00337585. PMID 7745322
- [Result] Iesalnieks I, Ommer A, Petersen S, Doll D, Herold A. German national guideline on the management of pilonidal disease. Langenbecks Arch Surg. 2016 Aug;401(5):599-609. doi: 10.1007/s00423-016-1463-7. Epub 2016 Jun 16. PMID 27311698
- [Result] Milone M, Velotti N, Manigrasso M, Anoldo P, Milone F, De Palma GD. Long-term follow-up for pilonidal sinus surgery: A review of literature with metanalysis. Surgeon. 2018 Oct;16(5):315-320. doi: 10.1016/j.surge.2018.03.009. Epub 2018 Apr 24. PMID 29699781
- [Result] Johnson EK, Vogel JD, Cowan ML, Feingold DL, Steele SR; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons' Clinical Practice Guidelines for the Management of Pilonidal Disease. Dis Colon Rectum. 2019 Feb;62(2):146-157. doi: 10.1097/DCR.0000000000001237. No abstract available. PMID 30640830